CLINICAL TRIAL: NCT01090479
Title: Efficacy of Home Pre-Operative Use of 2% Chlorhexidine Cloths Prior to Shoulder Surgery
Brief Title: Pre-operative Preparation Using 2% Chlorhexidine Cloth For Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Sage Products, Inc. (Industry)
Responsible Party: Principal Investigator, Gordon Nuber, Professor of Orthopaedics, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2% Chlorhexidine Cloths; NCT00829023 (obsolete NCT alias)
Record Dates: First submitted 2010-03-18; First posted 2010-03-22 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-04

CONDITIONS: Post-operative Surgical Site Infections
Keywords: Surgical site infections; Chlorhexidine; Shoulder surgery
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): This group will perform an ordinary shower the night prior and the morning of their scheduled surgery date.
- 2% Chlorhexidine cloth (Experimental): This group will use the 2% chlorhexidine wipes the night prior as well as the morning of their surgery date.
  Interventions: Drug: 2% Chlorhexidine cloth

INTERVENTIONS:
Drug: 2% Chlorhexidine cloth — The 2% Chlorhexidine cloth will be applied to the operative extremity the night prior and the the morning of their surgery.
  Arms: 2% Chlorhexidine cloth

SUMMARY:
We intend to determine how effective the use of a 2% Chlorhexidine Cloth is in terms of eliminating the bacterial load on patients undergoing shoulder surgery. We will be comparing the Chlorhexidine Cloths with a control group which will be performing an ordinary shower prior to surgery. At this time, it is standard of care to only take an ordinary shower the evening prior, and the morning of surgery.

DETAILED DESCRIPTION:
The use of home preoperative chlorhexidine wash has been used in various surgical fields for the prevention of perioperative infections. However, it's use in shoulder surgery has not been published up to this point. The shoulder has a unique microbial flora due to the prevalence of Propionibacterium acnes, a bacteria implicated in surgical site infections after shoulder surgery. This study is designed to examine the efficacy of using a preoperative Sage 2% chlorhexidine cloth in reducing bacterial load in the pre-operative area as well as in reducing post-operative surgical site infections after shoulder surgery. This study will compare the rate of post-operative infections and also the rate of positive skin cultures. The skin cultures will be obtained in the preoperative area from subjects who used the Sage 2% Chlorhexidine cloth protocol pre-operatively (n=50) versus those who used only soap and water (n=50).

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing shoulder surgery (open or arthroscopic)

Exclusion Criteria:

* Patient unwilling to comply with instructions
* Active infection in the operative extremity
* Documented allergic reaction to chlorhexidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Nuber, M.D., Principal Investigator — Professor of Orthopaedic Surgery
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Derived] Murray MR, Saltzman MD, Gryzlo SM, Terry MA, Woodward CC, Nuber GW. Efficacy of preoperative home use of 2% chlorhexidine gluconate cloth before shoulder surgery. J Shoulder Elbow Surg. 2011 Sep;20(6):928-33. doi: 10.1016/j.jse.2011.02.018. Epub 2011 May 25. PMID 21612945
- [Derived] Saltzman MD, Nuber GW, Gryzlo SM, Marecek GS, Koh JL. Efficacy of surgical preparation solutions in shoulder surgery. J Bone Joint Surg Am. 2009 Aug;91(8):1949-53. doi: 10.2106/JBJS.H.00768. PMID 19651954

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | 2% Chlorhexidine Cloth
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | 2% Chlorhexidine Cloth | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 43 | 89
  >=65 years | 4 | 7 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (8) | 49.0 (9) | 50.5 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 36 | 61
  Male | 25 | 14 | 39
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Clinically Diagnosed Infection
Time Frame: 2 months post-operatively
Measure: Number; unit: participants
Arm/Group | Control | Chlorhexidine
Number analyzed (Participants) | 50 | 50
participants | 0 | 0

2. Secondary Outcome: Qualitative and Quantitative Bacterial Cultures of the Operative Shoulder Just Prior to Surgery
Description: Rate of positive cultures from entire shoulder region (combined from axilla and posterior shoulder)
Time Frame: 7 days
Population: Rate of positive cultures from entire shoulder region (combined from axilla and posterior shoulder)
Measure: Number; unit: percentage of participants
Groups:
- Control: Soap and water
- Chlorhexidine: 2% chlorhexidine gluconate impregnated cloths
Arm/Group | Control | Chlorhexidine
Number analyzed (Participants) | 50 | 50
percentage of participants | 94 | 66

ADVERSE EVENTS:
Arm/Group | Control | 2% Chlorhexidine Cloth
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
No specific limitations other than the study was underpowered to detect a difference in the clinical infection rate between the chlorhexidine and control groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No